CLINICAL TRIAL: NCT02360046
Title: The Influence of Different Hydrocortisone Replacement Doses on the Partitioning and Flexibility of Ectopic Lipids (Intrahepatocellular IHCL and Intramyocellular IMCL) in Patients With Corticotropic Hypopituitarism, a Randomised Placebo-controlled Double-blind Trial
Brief Title: The Influence of Different Hydrocortisone Replacement Doses on the Partitioning and Flexibility of Ectopic Lipids in Patients With Corticotropic Hypopituitarism
Acronym: Hydrocort
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 211/14; 2014 DR 4137 (Other: Swissmedic)
Record Dates: First submitted 2015-01-16; First posted 2015-02-10 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Hypopituitarism; Hydrocortisone; Lipids; Fatty Acids, Nonesterified; Insulin Sensitivity
MeSH Terms: conditions — Hypopituitarism; Insulin Resistance | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Higher hydrocortisone dose (Other): Established hydrocortisone replacement therapy plus 10mg of hydrocortisone
  Interventions: Drug: Hydrocortisone
- Lower hydrocortisone dose (Other): Established hydrocortisone replacement therapy plus placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydrocortisone — Established Hydrocortisone replacement therapy plus Hydrocortisone (10mg/day)
  Arms: Higher hydrocortisone dose
Drug: Placebo — Established Hydrocortisone replacement therapy plus Placebo (0mg Hydrocortisone)
  Arms: Lower hydrocortisone dose

SUMMARY:
This study aims at assessing the effect of today's standard of hydrocortisone dosage versus previous hydrocortisone dosage on flexibility and partitioning of ectopic lipid depots (IMCL and IHCL) after a standardised fat load followed by a short-term aerobic exercise in patients with corticotropic pituitary insufficiency.

DETAILED DESCRIPTION:
Background

The investigators and others have shown that long-term hydrocortisone replacement therapy at higher doses of hydrocortisone replacement therapy at higher doses of hydrocortisone replacement (as previously recommended) is associated with higher mortality. The pathophysiology for the association of hydrocortisone-replacement dose and mortality remains unclear. A possible underlying mechanism is nonalcoholic fatty liver disease which is more prevalent in patients with hypopituitarism. Patients with non-alcoholic fatty liver disease are at a higher risk for overall-mortality.

It remains to be established whether the insulin resistance, associated with increased intrahepatocellular lipids and increased intramusculoskeletal lipids, is implicated in the pathophysiology of these epidemiological findings.

Interestingly, it has been shown that a reduction of hydrocortisone replacement dose from 20-30mg/d to 10-15mg/d resulted in a loss of body fat and a significant decrease of plasma total cholesterol and triglyceride concentration. The effect of IMCL and IHCL is so far unknown.

Patients with hypopituitarism with hydrocortisone replacement therapy provide a unique disease model to study the short-term effects of previously recommended dose (higher dose) of hydrocortisone versus lower dose of HC replacement therapy on ectopic lipids (IMCL; IHCL) lipids, as well as on subcutaneous and visceral fat mass and on parameters of insulin resistance. Combining MRI and MR-spectroscopy techniques, different fat mass (subcutaneous and visceral) and ectopic lipids can be repeatedly and non-invasively assessed.

Objective

To investigate the impact of today's standard of hydrocortisone dosage (lower) versus previous (higher) hydrocortisone dosage on flexibility and partitioning of ectopic lipid depots after a standardised fat load followed by a short-term aerobic exercise in patients with corticotropic pituitary insufficiency.

Methods

Ectopic lipids are measured by MR-spectroscopy, separate assessment of visceral and subcutaneous fat mass will be performed by MR-imaging, standardized exercise capacity test using spiroergometry. Short-time exercise consists of 2h aerobic cycling at 50% VO2max. Laboratory analysis include lipid profile, free fatty acids, HOMA-Index, hormones.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients
* Corticotropic pituitary insufficiency
* Capable to exercise during 120 minutes on a bicycle
* Normal ECG during ergometry

Exclusion Criteria

* Concomitant medication with NSAID, anticoagulants, digoxin, salbutamol, anticonvulsants, cholinesterase inhibitor, pancuronium
* Abnormal liver, renal or thyroid function, heart failure
* Hemophilia
* Diabetes mellitus
* Severe dyslipidemia
* Active neoplasia
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the study
* Lack of safe contraception
* Known or suspected non-compliance
* Drug or alcohol abuse
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the study
* Previous enrolment into current study
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Inability to exercise
* Contraindications to exposure to a 3 T magnetic field
* Major depression, psychosis, claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in flexibility of Intramyocellular Lipids (IMCL) Measured in mmol/L | 3 months
  Measured in mmol/L
Change from baseline in flexibility of Intrahepatocellular Lipids (IHCL) Measured in mmol/L | 3 months
  Measured in mmol/L

SECONDARY OUTCOMES:
Free Fatty Acids (FFA) availability during exercise before and after additional hydrocortisone/placebo Measured in mmol/L | At baseline, 3 months
  Measured in mmol/L
Flexibility of ectopic fat stores, defined as difference between intramyocellular/intrahepatocellular lipid concentration before and after exercise, and their possible relation to insulin sensitivity before and after additional hydrocortisone/placebo | At baseline, 3 months
Free Fatty Acids (FFA) availability during exercise and the possible relation to insulin sensitivity before and after additional hydrocortisone/placebo Measured in mmol/L | At baseline, 3 months
  Measured in mmol/L
Effect of exercise on insulin at baseline | At baseline
Effect of exercise on insulin at 3 months | 3 months
Effect of exercise on catecholamines at baseline | At baseline
Effect of exercise on catecholamines at 3 months | 3 months
Effect of exercise on growth hormone at baseline | At baseline
Effect of exercise on growth hormone at 3 months | 3 months
Effect of exercise on cortisol at baseline | At baseline
Effect of exercise on cortisol at 3 months | 3 months
Effect of exercise on lactate at baseline | At baseline
Effect of exercise on lactate at 3 months | 3 months
Effect of exercise on glucose at baseline | At baseline
Effect of exercise on glucose at 3 months | 3 months
Effect of exercise on inflammatory markers at baseline | At baseline
Effect of exercise on inflammatory markers at 3 months | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Christ, MD, PhD, Principal Investigator — Division of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Bern; Chris Boesch, MD, PhD, Principal Investigator — AMSM; Division of Radiology, University Hopsital of Bern, Inselspital
Locations (1):
- Division of Endocrinology, Diabetes and Clinical Nutrition, University Hospital Berne, Bern, Switzerland

REFERENCES:
- [Background] Boesch C, Slotboom J, Hoppeler H, Kreis R. In vivo determination of intra-myocellular lipids in human muscle by means of localized 1H-MR-spectroscopy. Magn Reson Med. 1997 Apr;37(4):484-93. doi: 10.1002/mrm.1910370403. PMID 9094069
- [Background] Danilowicz K, Bruno OD, Manavela M, Gomez RM, Barkan A. Correction of cortisol overreplacement ameliorates morbidities in patients with hypopituitarism: a pilot study. Pituitary. 2008;11(3):279-85. doi: 10.1007/s11102-008-0126-2. PMID 18459045